CLINICAL TRIAL: NCT07144865
Title: Effects of Anti-VEGF Agents on Angiogenic Factors in FVMs Impact of Anti-VEGF Therapy on Myofibroblast Products and Profibrotic Factors in FVMs Influence of Anti-VEGF Treatment on Pericyte Markers in FVMs
Brief Title: Biological Changes in Fibrovascular Membranes of Patients With Proliferative Diabetic Retinopathy Following Faricimab Injection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bojie Hu (Other)
Responsible Party: Sponsor-Investigator, Bojie Hu, Chief physician, Tianjin Medical University Eye Hospital
Organization: Tianjin Medical University Eye Hospital (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TianjinMUEHhbj100; Not provided (Other Grant/Funding Number: Bojie Hu); not provided (Other: Tianjin medical university eye hospital)
Record Dates: First submitted 2025-08-02; First posted 2025-08-28 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Proliferative Diabetic Retinopathy
MeSH Terms: interventions — KH902 fusion protein; faricimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Faricimab (IVF) (Active Comparator): Participants were randomly assigned to receive intravitreal injections of either faricimab (IVF, n=4) or conbercept (IVC, n=4) based on a randomisation protocol. To establish a baseline comparison, FVMs were obtained from three treatment-naive patients who served as controls. All participants underwent surgery 4 days after the intravitreal anti-VEGF injections.
  Interventions: Drug: Faricimab
- Conbercept (IVC) (Active Comparator): Participants were randomly assigned to receive intravitreal injections of either faricimab (IVF, n=4) or conbercept (IVC, n=4) based on a randomisation protocol. To establish a baseline comparison, FVMs were obtained from three treatment-naive patients who served as controls. All participants underwent surgery 4 days after the intravitreal anti-VEGF injections.
  Interventions: Drug: conbercept ophthalmic injection （0.5mg）

INTERVENTIONS:
Drug: conbercept ophthalmic injection （0.5mg） — Participants were randomly assigned to receive intravitreal injections of either faricimab (IVF, n=4) or conbercept (IVC, n=4) based on a randomisation protocol. To establish a baseline comparison, FVMs were obtained from three treatment-naive patients who served as controls. All participants underwent surgery 4 days after the intravitreal anti-VEGF injections.
  Other Names: conbercept
  Arms: Conbercept (IVC)
Drug: Faricimab — According to the randomization protocol, participants were randomly assigned to receive intravitreal injections of faricimab (IVF, n=4) or conbercept (IVC, n=4). To establish a baseline comparison, FVMs were obtained from three treatment-naïve patients as controls. All participants underwent surgery 4 days after intravitreal anti-VEGF injection.
  Arms: Faricimab (IVF)

SUMMARY:
DR is a common microvascular complication of DM that significantly impacts vision. Approximately one-third of DM patients develop DR, with 10% progressing to PDR. PDR is characterized by retinal ischemia-induced VEGF overexpression and pathological NV. NV proliferates along the vitreoretinal interface, potentially forming FVMs that increase RD risk and may lead to TRD.

FVM formation directly affects PPV complexity. Preoperative anti-VEGF injection reduces intraoperative bleeding and eliminates NV, but may accelerate fibrosis. Previous studies mainly focused on angiogenic/profibrotic factor changes in AH/VH, but whether FVM changes mirror these remains unclear.

This study compared mRNA levels of relevant factors in FVMs from PDR patients treated with faricimab versus conbercept, and investigated their effects on angiogenesis and fibrosis progression in FVMs.

DETAILED DESCRIPTION:
Diabetic retinopathy (DR) is one of the most common microvascular complications of diabetes that significantly affects the visual health of patients. The incidence of DR is increasing annually worldwide, with approximately one-third of patients with diabetes developing DR and approximately 10% progressing to proliferative diabetic retinopathy (PDR), which is an advanced stage of DR characterised primarily by retinal ischaemia that leads to the overexpression of vascular endothelial growth factor (VEGF) and the formation of abnormal neovascularization. These new blood vessels proliferate along the vitreoretinal interface, potentially resulting in the formation of fibrovascular membranes (FVM). The presence of FVM not only increases the risk of retinal detachment but may also lead to severe complications such as tractional retinal detachment (TRD).

The formation and characteristics of FVMs directly influence the complexity of pars plana vitrectomy (PPV). Preoperative injection of anti-vascular endothelial growth factor (anti-VEGF) agents is an effective strategy to reduce intraoperative bleeding and eliminate neovascularization (NV). However, per previous studies, anti-VEGF therapy may accelerate the progression of fibrosis. Changes in profibrotic factors in FVM have garnered significant interest. Previous studies have mainly focused on the changes in angiogenic and profibrotic factors in the aqueous humor or vitreous humor. However, whether the changes in these factors in the FVM are consistent with those in the vitreous and aqueous humors remains a question worth exploring.

In this study, researchers compared the mRNA levels of relevant factors in the FVMs of patients with PDR treated with faricimab or conbercept. Additionally, we investigated the effects of different anti-VEGF agents on the progression of angiogenesis and fibrosis in the FVMs of patients with PDR.

ELIGIBILITY:
Inclusion Criteria:

(1) Diagnosis of proliferative diabetic retinopathy; (2) no prior anti-VEGF treatment within three months; (3) presence of fibrovascular membrane; (4) without ocular or systemic comorbidities

Exclusion Criteria:

(1) history of prior vitrectomy; (2) presence of non-proliferative diabetic retinopathy; (3) coexisting systemic or ocular comorbidities, including, but not limited to, glaucoma, retinal vein occlusion, or rhegmatogenous retinal detachment; and (4) received anti-VEGF therapy within 3 months preceding enrolment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-04-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Concentration of Anti-VEGF Agents on Angiogenic Factors in FVMs | 4 days after injection
  VEGF ANG-2
Concentration of of Anti-VEGF Therapy on Myofibroblast Products and Profibrotic Factors in FVMs | Four days after the medication injection
  Fibronectin（FN1), connective tissue growth factor (CTGF), alpha-smooth muscle actin (α-SMA), and transforming growth factor beta (TGF-β)
Concentration of anti-VEGF treatment on pericyte markers in FVMs | Four days after the medication injection
  neural glial antigen 2 (NG2), and platelet derived growth factor receptor beta (PDGFR-β)

SECONDARY OUTCOMES:
Rate of Neovascularization on FVMs (SNV/SFVM, %) | 1, 2, 3, and 4 days after injection
  The areas of FVMs (SFVM) and neovascularization (SNV) were then calculated. The NV of the FVMs was quantified as the SNV/SFVM ratio (NV area to total FVM area).

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin medical university eye hosipital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No
Not considering it for the time being

REFERENCES:
- [Background] Takahashi N, Abe I, Kira S, Ishii Y. Role of epicardial adipose tissue in human atrial fibrillation. J Arrhythm. 2023 Feb 19;39(2):93-110. doi: 10.1002/joa3.12825. eCollection 2023 Apr. PMID 37021018
- [Background] Montero JA, Ruiz-Moreno JM, Correa ME. Intravitreal anti-VEGF drugs as adjuvant therapy in diabetic retinopathy surgery. Curr Diabetes Rev. 2011 May;7(3):176-84. doi: 10.2174/157339911795843104. PMID 21438852